CLINICAL TRIAL: NCT04074798
Title: Hyperventilation in Patients With Chronic Low Back Pain
Acronym: HELBP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: ZOL (Other)
Responsible Party: Principal Investigator, Lotte Janssens, Prof. dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CME ZOL - CTU2019078
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Low Back Pain, Recurrent; Hyperventilation Syndrome
MeSH Terms: conditions — Low Back Pain | interventions — Postural Balance

STUDY DESIGN:
Intervention Model Description: Patients with low back pain are compared to patients without low back pain (healthy controls).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with low back pain (Active Comparator)
  Interventions: Behavioral: assessment of hyperventilation, postural control and psychological behavior
- Healthy controls (Sham Comparator)
  Interventions: Behavioral: assessment of hyperventilation, postural control and psychological behavior

INTERVENTIONS:
Behavioral: assessment of hyperventilation, postural control and psychological behavior — assessment of hyperventilation, postural control and psychological behavior

SUMMARY:
Low back pain (LBP) is the leading cause of disability worldwide. Impaired postural control is a key factor in the development and maintenance of LBP. Moreover, the prevalence of LBP is associated with impairments in diaphragm function, symptoms of dyspnea, and dysfunctional breathing. However, the association between LBP (and more specifically postural control) and hyperventilation remains unknown. The main objective of this project is to investigate whether the presence of recurrent non-specific LBP is related to the presence of hyperventilation, when classified either objectively by decreased carbon dioxide values (demonstrating hypocapnia) or by symptoms while showing normal carbon dioxide values. Moreover, the investigators will explore whether psychosocial factors play a role in this relation. Subsequently, the investigators will examine whether hyperventilation in LBP patients is related to impaired postural control, and more specifically to a decreased postural contribution of the diaphragm.

ELIGIBILITY:
Inclusion Criteria Patients:

* Chronic primary low back pain (>12 weeks) as diagnosed by a medical doctor

Inclusion Criteria Healthy controls:

* No low back pain

Exclusion Criteria:

* Insufficient understanding of Dutch language
* Previous spinal surgery
* Chronic Obstructive Lung Disease, Interstitial Lung Disease, pulmonary vascular disease, asthma except for exertional asthma
* Acute cardiovascular or gastrointestinal disorders
* Neuromuscular disease interfering with normal lower limb or trunk functioning
* Acute pain or secondary chronic pain
* Pregnant and lactating women
* Major psychiatric conditions
* Acute lower limb problems
* Vestibular disorders

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Nijmegen questionnaire | Day 1
  Questionnaire evaluating hyperventilation symptoms, 16 items, total score range 0-64
Nijmegen questionnaire | Day 4
  Questionnaire evaluating hyperventilation symptoms, 16 items, total score range 0-64
PetCO2 | Day 1
  End-tidal carbon dioxide pressure measured with a capnograph
Postural control | Day 1
  upright standing balance measured by center of pressure by force plate

SECONDARY OUTCOMES:
Breathing frequency | Day 1
  amount of breaths per minute, inspiratory and expiratory time
Breathing pattern (abominal and thoracic) | Day 1
  abdominal or thoracic contribution to one breath measured by respiratory inductance plethysmography
Numerical Rating Scale for low back pain (NRS) | Day 1
  11 point Likert scale evaluating severity/intensity of back pain, ranging from 0 (no pain) to 11 (worst pain imaginable)
Oswestry Disability Index version 2.1a (ODI-2.1a) | Day 1
  Questionnaire evaluating disability. 10 items Total score range from 0-100
12-item Short form Health Survey (SF-12) | Day 1
  Questionnaire evaluating physical and mental components of health related quality of life. 12 items. Total score range 12-56.
Fear Avoidance Component Scale (FACS) | Day 1
  Questionnaire evaluating fear-avoidance related to pain. 20 items Total score range from 0-100
Tampa Scale for Kinesiophobia (TSK) | Day 1
  Questionnaire evaluating kinesiophobia related to pain. 17 items. Total score range from 17-68
Pain Catastrophizing Scale (PCS) | Day 1
  Questionnaire evaluating catastrophizing. 13 items, 5 point Likert scale. Total score 0-52
Need for Controllability and Predictability Questionnaire (NCP-Q) | Day 1
  Questionnaire evaluating the need for being able to control and predict situations. 15 items, 5 point Likert scale. Total score range 15 - 75
Positive And Negative Affect Schedule (PANAS) | Day 1
  Questionnaire evaluating positive and negative affect. 10 items positive affect, 10 items negative affect, 5 point Likert scale. Total score range per affect: 10 - 50
Pain Solutions Questionnaire (PaSoL) | Day 1
  Questionnaire evaluating assimilative and accommodative responses to problems associated with pain. 14 items, 7 point Likert scale. Total score range 0 - 84
Toronto Alexithymia Scale 20 (TAS-20) | Day 1
  Questionnaire evaluating characteristics linked to alexithymia. 20 items, 3 factors. Total score range 20 - 100
Interoceptive Awareness Questionnaire (IAQ) | Day 1
  Questionnaire evaluating adaptive and maladaptive body awareness. 19 items, 5 point Likert scale.
Fremantle Back Awareness Questionnaire (FreBAQ) | Day 1
  Questionnaire evaluating back specific perceptual awareness. 9 items, 5 point Likert scale. Total score range 0-36
Vragenlijst belastende ervaringen (VBE) - short version | Day 1
  Questionnaire evaluating aversive experiences in adult life. 11 items should be scored with yes or no. If yes a score on a 5 point Likert scale should be given.
Multidimensional Perfectionism Scale (MPS) | Day 1
  Questionnaire evaluating adaptive and maladaptive perfectionism. 35 items, 5 point Likert scale. Total score range 35 - 175
International Physical Activity Questionnaire - Short Form (IPAQ-SF) | Day 1
  Questionnaire evaluating subjective level of physical activity. 7 questions regarding amount of time spent on certain activities.

OTHER OUTCOMES:
Heart rate | Day 1
  ECG measurement to determine heart rate variability
Skin conductance | Day 1
  The resistance / conductance of the skin, stress physiological measure
Activity of abdominal muscles | Day 1
  The amount of muscle activation measured by electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Lotte Janssens, PhD, PT, Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No